CLINICAL TRIAL: NCT01230489
Title: The Efficacy of "MediHoney" to Facilitate Catheter Exit-Site Surgical Wound Healing and Prevention of Wound Bacterial Colonization: A Randomized, Open-label, Controlled, Clinical Trial
Brief Title: The Efficacy of "MediHoney" to Facilitate Catheter Exit-Site Surgical Wound Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Breakdown of communication between departments involved
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1171097
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-03

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): This group will undergo the current standard of care for post operative exit sites at the involved institutions. This group will act as the control or the group to which the interventional group will be compared too.
- MediHoney (Experimental): This study group will have the dry 2 x 2 dressing replaced with a honey 2 x 2 dressing. Additionally all indentations in the exit site wound will be filled with honey ointment prior to the application of the dressing.
  Interventions: Biological: MediHoney

INTERVENTIONS:
Biological: MediHoney — In this group a Medihoney 2 x 2 will be used in place of the standard dry 2 x 2 currently used as the wound dressing. Also all indentations of the wound will be filled with Medi-Honey ointment prior to the application of the dressing.
  Other Names: Honeycolloid Dressing; Leptospermum honey
  Arms: MediHoney

SUMMARY:
To evaluate the efficacy of honey as a post surgical exit site care process to promote healing and prevent infectious bacterial colonization of newly created exit sites. It has been shown in the medical literature that honey has properties that are conducive to healing and the prevention of infection. In one study it was demonstrated that in urethral injury in the rat treated with honey the injury healed with none of the usual formation of fibrous tissue seen in such healing processes, that there was no reduction in the luminal diameter usually seen, and that the cells lining the urethra were uncompromised in any way, i.e. totally normal and healthy. We feel that if an exit site can be healed quickly with good normal tissue being developed that the patient will have a much better chance to keep that exit healthy reducing time, cost, and disruption of lifestyle. Other positive aspects of honey are it has the low pH required for good healthy tissue healing, it works in the presence of wound fluids, and it has never been shown to produce a resistant bacterial strain.

DETAILED DESCRIPTION:
The exit site (ES) of any transcutaneous device, or foreign body, through the skin presents as the site most vulnerable in terms of device survival. With the large numbers of catheters in use in chronic dialysis today exit-site care for the prevention of infection is of critical importance in reducing morbidity and mortality. Pericatheter infection is the number one cause of catheter loss in peritoneal dialysis patients.

It appears that honey is a compound with a multi-factorial mode of action. It is thought that with most honeys, the antimicrobial action stems from its high osmolality and the fact that it produces continuous non-cytotoxic levels of hydrogen peroxide due to enzymatic break down of the sugar. Honey also has a low pH which is not conducive for most bacterial growth but is good for wound healing.

Observational reports have shown some success in healing infected wounds, ulcers, protection of plastic surgery transplants, burns, herpetic skin lesions, and atopic dermatitis. Honey has also been shown to have antimicrobial action against a broad spectrum of fungi and bacteria including antibiotic resistant bacteria. Another study reports that honey reduces inflammation, edema, and promotes angiogenesis.

In an animal study of urethral injury it was shown that contrary to controls, there was a total healing with restoration of normal urethral epithelium and connective tissue with complete absence of fibrosis and inflammation. There was also no narrowing of the lumen as seen in the other study groups.

A study of prophylactic exit-site care of hemodialysis catheters comparing honey and Mupirocin demonstrated that results with honey were comparable to that of Mupirocin. However, unlike Mupirocin, there has not been an emergence of honey-resistant bacterial strains which makes it an attractive alternative agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring dialysis due to loss of kidney function
* Patients choosing Peritoneal Dialysis (PD) for treatment
* All PD patients having an indwelling PD catheter placed

Exclusion Criteria:

* Patients younger than 18 years of age
* Prisoners
* Patients with mental defect
* Veteran Administration patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold L Moore, MA, Principal Investigator — University of Missouri, School of Medicine, Department of Medicine
Locations (1):
- University of Missouri Department of Medicine; Dialysis Clinic, Inc., Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 participants were recruited from surgical clinics.
Pre-assignment Details: Data is unavailable as no analysis has occurred. The study was terminated to due loss of communication between the surgical and research departments.
Groups:
- Surgical Catheter Dressings: Participants were randomized to receive either a standard of care dressing to their surgical wound catheter exit site or the MediHoney dressing.
  Data is unavailable as no analysis has occurred. The study was terminated to due loss of communication between the surgical and research departments.
Period: Overall Study
Arm/Group | Surgical Catheter Dressings
Started | 13
Completed | 8
Not Completed | 5
Not completed — Death | 2
Not completed — Adverse Event | 2
Not completed — Treatment modality changed | 1

BASELINE CHARACTERISTICS:
Population: Participants were assigned to receive the standard care dressing or the MediHoney dressing. It is unknown how many were assigned to each arm due to research staff no longer being available.
Groups:
- Surgical Catheter Dressings: Participants randomized to either standard of care dressings or Medihoney dressings to catheter exit sites. The numbers allocated to each arm is unknown. Data is unavailable as no analysis has occurred. The study was terminated to due loss of communication between the surgical and research departments.
Arm/Group | Surgical Catheter Dressings
Number analyzed (Participants) | 13
Age, Customized [Count of Participants; unit: Participants]
  Age 18 - 90 years | 13
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Unknown | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Time From Catheter Implantation to First Exit Site Infection.
Description: The outcome measure is the length of time from implantation until the patient has first exit site infection or two years which ever is shortest.
Time Frame: Two years
Population: Data is unavailable as no analysis has occurred. The study was terminated to due loss of communication between the surgical and research departments.
Groups:
- Surgical Catheter Dressings: Participants randomized to either standard of care dressings or Medihoney dressings to catheter exit sites.It is not known how many were assigned to each arm.
Arm/Group | Surgical Catheter Dressings
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Surgical Catheter Dressings: Participants randomized to either standard of care dressings or Medihoney dressings to catheter exit sites. Data is unavailable as no analysis has occurred. The study was terminated to due loss of communication between the surgical and research departments.
Arm/Group | Surgical Catheter Dressings
All-Cause Mortality (participants affected / at risk) | 2/13
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Catheter Dressings (N=13)
Perforated bowel (Gastrointestinal disorders) | 1 (1)
Yeast Infection (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No